CLINICAL TRIAL: NCT06379763
Title: Effect of Adding Diaphragmatic Breathing Exercise to Conventional Physiotherapy Intervention on Pain and Sleep Quality in Individuals With Non-specific Chronic Neck Pain: A Randomized Control Trial
Brief Title: Effect of Diaphragmatic Breathing Exercise on Pain and Sleep Quality in Individuals With Non-specific Chronic Neck Pain: A Randomized Control Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Islam Mazen Kamal Alnaqeeb, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 170/2024
Record Dates: First submitted 2024-04-07; First posted 2024-04-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Non-specific Chronic Neck Pain; Diaphragmatic Breathing Exercise
Keywords: diaphragmatic breathing; sleep Quality; pain; physiotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Pain

STUDY DESIGN:
Intervention Model Description: randomized clinical trial (RCT) Participants will be randomly allocated into two groups using the block randomization method. The following groups will be formed: experimental group A (diaphragmatic breathing plus conservative physiotherapy intervention, cervical neck ROM, neck stretching exercises), and group B,
Who Masked: Participant
Masking Description: the participants will not know which of exercises that will be giving for them more better in experimental or control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group one (Experimental): diaphragmatic breathing exercise in addition to conventional physiotherapy such as ROM, stretching exercises for superficial neck muscles
  Interventions: Other: diaphragmatic breathing exercise; Other: conventional physiotherapy exercise
- group two (Active Comparator): conventional physiotherapy exercise such as ROM, stretching exercises for superficial neck muscles
  Interventions: Other: conventional physiotherapy exercise

INTERVENTIONS:
Other: diaphragmatic breathing exercise — 15-minute diaphragmatic breathing exercise from a semi-Fowler's position. Patients will be instructed to position one hand on the chest and the other on the belly, gradually inhaling deeply through the nose, moving from functional residual capacity to total lung capacity, and holding the breath for three seconds. Patients will be advised to relax their shoulders, maintain quiet upper chest movement, and allow the abdomen to slightly rise. Subsequently, patients will exhale slowly through the mouth for up to five seconds. Diaphragmatic breathing exercises will be organized into three sets lasting 15 minutes, with 3 minutes of active exercise and a 2-minute rest period between sets. During rest intervals, patients will be instructed to breathe normally. If individuals experience dizziness or discomfort, the session will stop.
  Other Names: abdominal breathing exercise
  Arms: group one
Other: conventional physiotherapy exercise — conventional physiotherapy exercise such as ROM, stretching exercises for superficial neck muscles

SUMMARY:
This research focuses on adding diaphragmatic breathing to conventional physiotherapy sessions, particularly for patients suffering from chronic neck pain aged between 20-40 years in Jordan. Chronic neck pain is recognized as one of the most prevalent musculoskeletal pain disorders, significantly impacting physical, social, and psychological aspects of life. This issue leads to a decline in functional performance and work productivity, negatively affecting both individual and societal levels. Several factors, such as poor posture and prolonged use of smartphones, contribute to the exacerbation of non-specific chronic neck pain. These problems also affect respiratory muscles, particularly the diaphragm responsible for primary respiration, resulting in a shift from abdominal to chest breathing. This alteration increases the use of neck muscles, subsequently intensifying neck pain and negatively impacting sleep quality in these individuals. The primary objective of this therapeutic study is to investigate the role of adding diaphragmatic breathing to physiotherapy sessions in alleviating pain and improving sleep quality.

RCT study will investigate the effect of adding the diaphragmatic breathing to conventional physiotherapy treatment on pain and sleep quality over one month.

DETAILED DESCRIPTION:
Non-specific chronic neck pain (NSCNP) is discomfort originating in the area between the superior nuchal line and the spinous process of the initial thoracic vertebra, extending to the scapula region, anterior chest wall, head, or upper limb . NSCNP is defined as neck discomfort persisting for over 12 weeks and is categorized as mechanical neck pain . demonstrated that NSCNP is associated with factors like forward head posture and rounded shoulders. Prolonged smartphone use, exceeding 10 hours per week, is linked to neck pain development . Additionally, found a positive correlation between mobile phone use duration and neck pain intensity, suggesting that individuals with poor posture, spending more than 10 hours daily on their phones, increase activation of neck muscles, including superficial muscles like sternocleidomastoid, anterior scalene, and trapezius. Recent findings reported that 54% of participants used their phones for more than 4 hours daily, increasing the occurrence of NSCNP .

Several negative factors affect individuals with non-specific chronic neck pain, such as poor posture, prolonged use of mobile phones throughout the day, and unhealthy sleep habits, contributing to increased neck pain and disrupting normal breathing patterns. Therefore, incorporating simple breathing re-education exercises, such as diaphragmatic breathing, into conventional physiotherapy interventions is considered effective and beneficial. It is also time-efficient and cost-effective. Moreover, this exercise is easily performed in various situations.

The aim of this study

Primary aim:

To assess the effectiveness of adding diaphragmatic breathing exercise to conservative physiotherapy interventions on pain and sleep quality in individuals with non-specific chronic neck pain.

The research question for this study Does adding diaphragmatic breathing to conservative physiotherapy interventions decrease pain and improve sleep quality in individuals with non-specific chronic neck pain?

Methodology

* Study design This study will be a randomized clinical trial (RCT) conducted over four weeks, with two sessions per week.
* Recruitment procedures A total of 40 participants will be recruited through flyers at the University of Jordan and posters on social media. Participants who meet the inclusion criteria will be eligible to participate in this study. The researcher will explain the aim and methods of the study to each participant, and informed consent will be obtained before conducting the study. Participants who agree to participate will sign the consent form. Additionally, the researcher will inform participants that they are free to withdraw from the study at any time without facing any negative consequences.
* Inclusion criteria Participants aged between 20 and 40 who have experienced neck pain for more than 3 months will be included in the study.
* Exclusion criteria Individuals with neurological or cardiorespiratory problems, cancer, officially diagnosed sleep disturbances, or those experiencing neck pain for less than 3 months will be excluded from the study. Participants with psychological diseases will also be excluded.
* Randomization procedures Participants will be randomly allocated into two groups using the block randomization method. The following groups will be formed: experimental group A (diaphragmatic breathing plus conservative physiotherapy intervention, cervical neck ROM, neck stretching exercises), and group B, which will receive conventional physiotherapy, including simple neck ROM and neck stretching exercises. A random number generator will be used to generate a random sequence of numbers, available at https://www.randomizer.org/The experimental group will be allocated to odd numbers, and the control group will be allocated to even numbers. The group label will be placed in an envelope, sealed, and stacked according to the sequence generated by the random number generator. To ensure an equal distribution of males and females in each group, block randomization will be applied. In each block, consisting of four envelopes, two will be assigned for females and two for males. Accordingly, the random number generator will be utilized twice, generating numbers from 1 to 20 for females and 1 to 20 for males.
* Demographic data Demographic information to be collected will include age, gender, weight, height, type of work (profession), such as student, housewife, or office worker, marital status, use of medications, and smoking status (smoker or non-smoker).
* Outcoms Primary outcome measure (pain) will be assessed by both VAS, NDI The Visual Analog Scale (VAS) The Visual Analog Scale (VAS) will be used to assess pain intensity, ranging from 0 to 10, where 10 represents the highest degree of pain intensity . This scale has demonstrated good psychometric properties for use in chronic neck pain . Patients will be instructed to indicate the point on the 10-point scale that best represents the intensity of their pain. Pain levels will be assessed before and after the sessions.

The Neck Disability Index (NDI) The Neck Disability Index (NDI) is a self-reported scale comprising ten items, each evaluating distinct complaints related to neck pain, mainly focusing on limitations in daily activities. It is considered a valid and reliable tool for assessing the impact of neck pain on patients' functional activities. The ten questions cover pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each item is scored from 0 (no disability) to 5 (total disability), with a maximum possible score of 50. It takes approximately 5 minutes for patients to complete it. Additionally, the Arabic version of the Neck Disability Index will be used to assess pain before and after the sessions . This Arabic version has been revealed to be a reliable, valid, and responsive tool .

• Secondary outcome measure (sleep quality) The Pittsburgh Sleep Quality Index (PSQI) The Pittsburgh Sleep Quality Index (PSQI) is the most commonly used standardized questionnaire for the comprehensive assessment of sleep quality, developed by . It can differentiate between good and poor sleepers and the questionnaire consists of 19 self-reported items, each categorized into one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Additionally, for clinical purposes, five extra questions rated by the respondent's roommate or bed partner are included, but they are not scored. Clinicians assess these components when individuals report sleep complaints. The definition of poor sleep varied between studies, with a cutoff PSQI global score ranging from 5 to 8 . This questionnaire will be used to assess sleep quality both before and after treatment.

additionally, The estimation of the sample size was performed using G*Power for a two-group design involving two repeated measures (pre and post) in a two-tailed test. To achieve a statistical power of 0.80 with an alpha level set at 0.05 and a medium effect size of f-test = 0.25, we took into consideration a dropout rate of 20%. Thus, the sample size is estimated to be around 40.

Intervention Eight treatment sessions will be conducted for all participants individually in a suitable environment.

Experimental group: Participants in this group will undergo a 15-minute of simple cervical neck range of motion (ROM) exercises, followed by stretching exercises for superficial neck muscles (sternocleidomastoids, upper trapezius, anterior scaleni) (3-5 times, 30-sec holds for each muscle). This will be followed by a 15-minute diaphragmatic breathing exercise from a semi-Fowler's position. Patients will be instructed to position one hand on the chest and the other on the belly, gradually inhaling deeply through the nose, moving from functional residual capacity to total lung capacity, and holding the breath for three seconds. Patients will be advised to relax their shoulders, maintain quiet upper chest movement, and allow the abdomen to slightly rise. Subsequently, patients will exhale slowly through the mouth for up to five seconds. Diaphragmatic breathing exercises will be organized into three sets lasting 15 minutes, with 3 minutes of active exercise and a 2-minute rest period between sets. During rest intervals, patients will be instructed to breathe normally. If individuals experience dizziness or discomfort, the session will stop. Each session will last for 30 minutes, and the diaphragmatic breathing exercises require a high concentration and a calm environment, so they will be conducted in a suitable environment.

Control group: Participants in this group will undergo a 15-minute of stretching and ROM exercises, including simple cervical neck ROM for 5 minutes and stretching exercises for superficial neck muscles (sternocleidomastoids, upper trapezius, anterior scaleni) for 10 minutes (3-5 times, 30-sec holds for each muscle).

Home exercise: All participants will be assigned home exercises to be performed once a week, consisting of two 5-minute postural exercises: stretching exercises for the pectoralis muscle and strengthening the rhomboids muscle through scapular squeezes. Additionally, participants in the experimental group will be provided with a 3-minute diaphragmatic breathing session. Each week, participants will fill out a checklist, and they will receive SMS reminders to enhance adherence. Furthermore, specific videos will be sent to increase their awareness about the importance of postural corrections and improving general health.

Data analysis:

Baseline data will be analyzed using descriptive statistics, displaying means, standard deviation, and frequencies. Additionally, the mixed analysis of variance (ANOVA) model will be employed to analyze the dependent variables, including the Neck Disability Index and sleep quality. This approach will help address the primary research questions. The statistically significant level will be set at p < 0.05. The data will be analyzed using SPSS 27.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 20 and 40
* experienced neck pain for more than 3 months

Exclusion Criteria:

* Individuals with neurological or cardiorespiratory problems
* Individuals with cancer
* Individuals with officially diagnosed sleep disturbances
* Individuals with experiencing neck pain for less than 3 months
* Individuals with psychological diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
neck pain | assessed before and after 4 weeks
  assessed by visual analogue scale. from 0 to 10 therefor 0 mean no pain where as 10 mean extremely pain
neck pain | assessed before and after 4 weeks
  assessed by neck disability index. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. The test can be interpreted as a raw score from 0 to 50, with a maximum score of 50, or as a percentage , therefor 0 mean no pain where as 50 mean extremely pain .

SECONDARY OUTCOMES:
sleep quality | assessed before and after 4 weeks
  assessed by The Pittsburgh Sleep Quality Index (PSQI). Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances. referred to as the global PSQI score, which ranges from 0 to 21. Zero mean good sleep quality Whereas Higher scores mean poor quality sleep

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No